CLINICAL TRIAL: NCT01581944
Title: Phase 3 Study of Experience With a Gonadotropin-releasing Hormone Agonist Prior to Myomectomy - Comparison of 2 Versus 3 Monthly Doses.
Brief Title: Gonadotropin-releasing Hormone Agonist Prior to Myomectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mt. Hope Maternity Hospital (Other)
Responsible Party: Principal Investigator, Dr. Bharat Bassaw, Senior Lecturer, Consultant, Head of Obstetrics and Gynaecology, Mt. Hope Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MtHopeMaternity0075
Record Dates: First submitted 2012-04-17; First posted 2012-04-20 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Fibroids
Keywords: myomectomy; GnRH; blood loss
MeSH Terms: conditions — Leiomyoma; Hemorrhage | interventions — Goserelin; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No Treatment (Control) (No Intervention): Women were randomised to receive no gonadotropin-releasing hormone agonist prior to myomectomy.
- 2 Doses Goserelin (Experimental): Women were randomised to receive 2 doses of 3.6mg of gonadotropin releasing hormone agonist prior to the myomectomy.
  Interventions: Drug: 2 Doses Goserelin
- 3 Doses Goserelin (Experimental): Women were randomised to receive 3 doses of the gonadotropin-releasing agonist (3.6mg monthly injections).
  Interventions: Drug: 3 Doses Goserelin

INTERVENTIONS:
Drug: 2 Doses Goserelin — 3.6mg administered monthly for 2 months prior to myomectomy
  Other Names: Gonadotropin Releasing Hormone Agonist
  Arms: 2 Doses Goserelin
Drug: 3 Doses Goserelin — 3.6mg administered monthly for 3 months prior to myomectomy
  Other Names: Gonadotropin Releasing Hormone Agonist
  Arms: 3 Doses Goserelin

SUMMARY:
Fibroids are common in the West Indian population (30-40% of reproductive women).Fibroids are benign growth in the womb or uterus and in order to preserve the fertility of women they, require an operation called myomectomy or shelling out of the fibroid. This procedure can be associated with large blood loss.

In current practice some obstetricians use a gonadotropin releasing hormone agonist prior to the operation to reduce blood loss. Gonadotropin releasing hormone agonist is used in current gynaecological practice to treat women with heavy periods.

In this study the investigators randomised women to either 2 or 3 doses of the gonadotropin agonist prior to their operation and no treatment. The intraoperative blood loss was measured. The study hypothesis: To determine whether administration of gonadotropin releasing hormone agonist prior to myomectomy reduces intraoperative blood loss.

DETAILED DESCRIPTION:
Variables noted preoperatively:

* Age
* Parity
* Ethnicity
* Ultrasound findings

Variables noted intra-operatively:

* Size of largest fibroid
* Estimated blood loss

ELIGIBILITY:
Inclusion Criteria:

* Women between the age of 20 and 45
* Symptomatic fibroids
* Presence of regular menstrual cycles
* Ultrasound confirmation of fibroids
* Normal cervical smear

Exclusion Criteria:

* Pregnancy
* The length of hospital stay was calculated in number of days from the date of the to the date of discharge
* Presence of endometriosis Previous myomectomy Ovarian, uterine or cervical malignancy female factor for subfertility

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss | 3 months
  Gonadotropin releasing hormone agonist Goserelin 3.6mg was administered for either 2 or 3 months prior to the operation.

SECONDARY OUTCOMES:
Blood transfusion requirement | Intraoperatively and in the postoperative period
  The hemoglobin level of each woman was measured on day 1 post operative and a blood transfusion was recommended if the hemoglobin level was <9g/dl.
The level of difficulty in enucleation of the fibroid and in achieving hemostasis. | Immediately after the operation
  The surgeons were asked to record the level of difficulty in enucleation (shelling out) of the fibroids and in securing hemostasis. They were asked to state if it was Easy, moderate or difficult.
Length of operation | Immediately after operation
  The length of operation was calculated from the skin incision to closure (minutes).
Length of hospital stay | Number of days from operation date to discharge date
  The length of hospital stay was calculated in number of days from the date of the to the date of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Bharat Bassaw, MBBS FRCOG, Principal Investigator — Mt. Hope Maternity Hospital
Locations (1):
- Gynaecological Outpatient Clinic; Mt. Hope Maternity Hospital, Champs Fleurs, Trinidad and Tobago